CLINICAL TRIAL: NCT05405283
Title: Randomized, Single-blinded, Multicenter Trial Comparing the Immune Response to a 2nd Booster Dose of COVID-19 mRNA Vaccine (Pfizer-BioNTech) or Sanofi /GSK B.1.351 Adjuvanted Vaccine in Adults Who Received 2 Doses of Pfizer-BioNTech mRNA Vaccine and a Booster Dose of Pfizer-BioNTech or Moderna mRNA Vaccine
Brief Title: Randomized, Single-blinded, Multicenter Trial Comparing the Immune Response to a 2nd Booster Dose of COVID-19 mRNA Vaccine (Pfizer-BioNTech) or Sanofi /GSK B.1.351 Adjuvanted Vaccine in Adults
Acronym: COVIBOOSTAnci1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: IREIVAC/COVIREIVAC Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AP211184; 2021-004550-33 (EudraCT Number)
Record Dates: First submitted 2022-06-03; First posted 2022-06-06 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Vaccines
Keywords: COVID 19; mRNA vaccines; Immunology; Sub-unit vaccine; Second booster
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comirnaty® (Pfizer-BioNTech) (Active Comparator)
  Interventions: Biological: 2nd booster with Comirnaty® (Pfizer-BioNTech)
- CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK (Experimental)
  Interventions: Biological: CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK

INTERVENTIONS:
Biological: 2nd booster with Comirnaty® (Pfizer-BioNTech) — In participants previously vaccinated with 3 doses of mRNA vaccine, he/she will receive one dose of Comirnaty® (Pfizer-BioNTech) vaccine as a second booster
  Arms: Comirnaty® (Pfizer-BioNTech)
Biological: CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK — In participants previously vaccinated with 3 doses of mRNA vaccine, he/she will receive one dose of CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK vaccine as a second booster
  Arms: CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK

SUMMARY:
The effectiveness of COVID-19 vaccines in reducing the risk of severe COVID-19 is currently demonstrated. In France, since the beginning of the vaccination campaign, 54,266,859 people have received at least one injection (ie. 80.5% of the total population), 53,354,698 people now have a complete vaccination schedule (ie. 79.1% of the total population) and since the beginning of the booster campaign, 39,558,416 people have received a 1st booster dose.

However, the data currently available on the persistence of immunity on the one hand, and the appearance of viral variants with reduced sensitivity to vaccine immunity on the other, suggest the need to administer booster doses at variable intervals depending on age and comorbidities. Real-life efficacy data from France and around the World confirm that people who have received a booster dose are better protected than those who have only received a primary vaccination schedule (HAS).

In this context, the Ministry of Health, has pronounced on the possibility of administering a second booster dose for people aged 60 and over. Moreover, the recommendations for the Haute Autorité de Santé for the 2nd booster dose in general population should be available in June 2022.

Three vaccines, mRNA BNT162b2 vaccine, Sanofi/GSK monovalent D614 and B.1.351 formulations were administered as 1st booster in the CoviBOOST trial. All three vaccines boosted antibodies and neutralizing response after a BNT162b2 initial course. Heterologous boosting with the Sanofi/GSK SARS-CoV-2 recombinant adjuvanted protein vaccine B.1.351 (Beta formulation) provided higher rates of neutralizing antibodies against variants, including Omicron BA.1, compared with the mRNA BNT162b2 vaccine. Due to the start of the study after the beginning of booster vaccination campaign in elderly, the enrollment of participants over 65 years of age was difficult so, only 8 subjects aged 60 years and over were enrolled. As vaccine immunogenicity is lower in older populations and is waning more rapidly, it is important to evaluate the adjuvanted vaccine in this population.

The objective of this ancillary study is to compare, in participants aged of 60 years and older and previously vaccinated with 3 doses of mRNA vaccine (2 doses of Pfizer BioNTech) and a 3rd dose of Pfizer BioNTech or Moderna, the immunogenicity of a second booster dose of the B.1.351 strain recombinant protein- based subunit vaccine to BNT162b2 (mRNA Pfizer BioNTech Vaccine).These results will provide important information for booster vaccination recommendations in this age group.

DETAILED DESCRIPTION:
The data currently available on the persistence of immunity on the one hand, and the appearance of viral variants with reduced sensitivity to vaccine immunity on the other, suggest the need to administer booster doses at variable intervals depending on age and comorbidities. Real-life efficacy data from France and around the World confirm that people who have received a booster dose are better protected than those who have only received a primary vaccination schedule (HAS).

Currently available data from the United States and the United Kingdom show that the protection conferred by the first booster dose diminishes after 3 months, particularly in persons 60 years of age and older, and justified the recommendation of a second booster dose.

Data from Israel show that a second booster dose (4th dose) reduces the rate of confirmed infections by a factor of 2 and the rate of severe disease by a factor of 4. The safety data, although limited, are reassuring.

In this context, the Ministry of Health, has pronounced on the possibility of administering a second booster dose for people aged 60 and over. Moreover, the recommendations for the Haute Autorité de Santé for the 2nd booster dose in general population should be available in June 2022.

The vaccines currently recommended in France, for booster vaccination are mRNA vaccines. However, some vaccines that were developed later in the clinic could present an interesting alternative in terms of reactogenicity, accessibility, cost and acceptability. Moreover, a heterologous vaccination scheme could be more immunogenic than a homologous scheme. Therefore, it is important to be able to evaluate these vaccines as a second booster dose.

The COVID 19 vaccines developed by Sanofi are based on a classical adjuvanted recombinant protein approach. Three candidate vaccines are under development, one based on the Spike protein of the SARS CoV-2 D614 strain, the other on the B.1.351 strain, and the third is a vaccine combining the two.

Three vaccines, mRNA BNT162b2 vaccine, Sanofi/GSK monovalent D614 and B.1.351 formulations were administered as 1st booster in the CoviBOOST trial. All three vaccines boosted antibodies and neutralizing response after a BNT162b2 initial course. Heterologous boosting with the Sanofi/GSK SARS-CoV-2 recombinant adjuvanted protein vaccine B.1.351 (Beta formulation) provided higher rates of neutralizing antibodies against variants, including Omicron BA.1, compared with the mRNA BNT162b2 vaccine.

Due to the start of the study after the beginning of booster vaccination campaign in elderly, the enrollment of participants over 65 years of age was difficult so, only 8 subjects aged 60 years and over were enrolled. As vaccine immunogenicity is lower in older populations and is waning more rapidly, it is important to evaluate the adjuvanted vaccine in this population.

The objective of this ancillary study is to compare, in participants aged of 60 years and older and previously vaccinated with 3 doses of mRNA vaccine (2 doses of Pfizer BioNTech) and a 3rd dose of Pfizer BioNTech or Moderna, the immunogenicity of a second booster dose of the B.1.351 strain recombinant protein- based subunit vaccine to BNT162b2 (mRNA Pfizer BioNTech Vaccine).These results will provide important information for booster vaccination recommendations in this age.

Participants enrolled will be healthy adults of 60 years old and over they will be recruited in 15 centers in mainland France, via the COVIREIVAC network.

The study will be a randomized, single-blinded, multicentre trial with two parallel arms:

ARM 1 receiving Pfizer-BioNTech vaccine

* Group 1.A: 1rst booster Pfizer
* Group 1.B: 1rst booster Moderna

ARM 2 receiving SP/GSK subunit B.1.351 vaccine

* Group 2.A: 1rst booster Pfizer
* Group 2.B: 1rst booster Moderna

Participants will undergo 4 visits :

* V1 (D0): inclusion, randomization, pregnancy test, PCR test, blood draw and administration of the booster dose
* V2 (D15): follow-up visit with a review of solicited and unsolicited local and systemic reactions that occurred since the last visit, and blood draw
* V3 (D28): follow-up visit with review of potential adverse events and blood draw
* V4 (D90): follow-up visit with review of potential adverse events and blood draw
* V4 (D180): follow-up visit with review of potential adverse events and blood draw

Blood samples will be used to conduct immunological analyses, and cellular analyses for a sub-category of 25 participants per group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years.
2. Adult in good health or with a stable health status if pre-existing medical history. Stable health status is defined as an existing disease that has not required a significant change in treatment or hospitalisation for worsening in the 3 months prior to inclusion, and for which no significant change in treatment or hospitalisation for worsening of the disease is envisaged in the near future.
3. For participants over 60 years of age who participated in Coviboost, to have received a booster dose of mRNA vaccine (Pfizer-BioNTech) administered at least 6 months before the 2nd booster dose
4. Not included in Coviboost (new participants to be recruited) and having received 2 doses of mRNA vaccine (Pfizer-BioNTech) with an interval of 3 to 6 weeks and a 1st booster dose of mRNA vaccine (Pfizer-BioNTech) or Moderna administered at least 6 months before the 2nd booster dose
5. Understands and agrees to comply with the study procedures.
6. Written informed consent signed by the participant and the investigator.
7. Person affiliated to a social security scheme.

Exclusion Criteria:

1. Acute febrile infection (body Acute febrile infection (body temperature ≥ 38.0°C) within the previous 72 hours and/or had symptoms suggestive of COVID-19 within the last 28 days or had case contact within the last 10 days before the inclusion visit.
2. Virologically documented (PCR or serology) history of COVID 19.
3. Immunosuppressive drugs such as corticosteroids at a dosage > 10 mg prednisone equivalent/day (excluding topical preparations and inhalers) within 3 months prior to inclusion or within 6 months for chemotherapies.
4. Treated with immunoglobulin or other blood product within 3 months prior to inclusion or scheduled for administration of immunoglobulin or blood product before the end of the study.
5. Known HIV, HCV or HBV infection.
6. Any condition, such as cancer, that may reduce the immune response.
7. Use of experimental Ig, experimental monoclonal antibodies or convalescent serum is not allowed during the study.
8. History of severe adverse reactions after vaccine administration including anaphylactic reaction and associated symptoms such as rash, difficulty breathing, angioedema and abdominal pain, or a history of an allergic reaction that may be exacerbated by a component of the SARS-COV-2 vaccine during the first vaccine injection.
9. Participant having been vaccinated against BCG in the previous year.
10. Having received a vaccination within 2 weeks prior to the 2nd booster dose or scheduled to receive a licensed vaccine 2 weeks after the 2nd booster dose.
11. Any bleeding disorder considered as a contraindication to an intramuscular injection, previous phlebotomy or receipt of anticoagulants.
12. Participation in other research involving humans (French classification Jardé 1 or Jardé 2) within 4 weeks prior to the inclusion visit, or participation in any other vaccine trial.
13. Subject under legal protection (e.g. guardianship, tutorship).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of a second booster 15 days after receiving the second booster | 15 days after second booster
  Proportion of patient with an increase of at least 10-fold between D0 and D15 after the 2nd booster dose in neutralizing antibody titers against SARS-CoV-2 D614,B.1.351, Delta and Omicron BA.1 and BA.2 viral strains, measured by a microneutralization technique.
  A 10-fold increase implies that the second titer is at least 2 dilutions higher than the first, which represents an unambiguous increase according to the state of the art of serum neutralization.

SECONDARY OUTCOMES:
Rate of neutralizing antibody titer against SARS-CoV-2 viral at 6 and 12 months | Up to 12 months after second booster
  The rate of neutralizing antibody titer against SARS-CoV-2 viral strains D614, Beta, Delta and Omicron BA.1 and BA.2, measured by microneutralization, until 6 months after the 2nd dose in each group.
Number and intensity of local and systemic adverse events at 28 days | Up to 28 days after second booster
  Number and intensity of local and systemic adverse events of any degree occurring up to day 7 after administration of the 2nd booster dose (assessed from the list of solicited adverse events); number and intensity of unsolicited local and systemic clinical events up to 28 days
Anti-Spike and anti-RBD IgG levels at 6 and 12 months | Up to 12 months after second booster
  Anti-Spike and anti-RBD IgG levels expressed as BAU/ml, according to WHO recommendations, at D15, D28, M3 and M6 after administration of the 2nd booster dose of mRNA vaccine vs. the 2nd dose of adjuvanted subunit B.1.351 vaccine;
Difference in anti-Spike and anti-RBD B.1.351 IgG level at 6 months and 12 months | 6 months
  Difference in anti-Spike and anti-RBD B.1.351 IgG levels between M3, M6 and M12
Difference in anti-Spike and anti-RBD B.1.351 IgG level at D15 | 15 days
  Difference in anti-Spike and anti-RBD B.1.351 IgG levels between D15 and D0
ELISPOT IFN CD4 and CD8 response | 15 days
  ELISPOT IFN CD4 and CD8 response at D15
Activated (CD71+) spike Beta specific B cells will also be sorted and cultured in single cells for further analysis of their BCR and their relationship with the early CSA response | Day 0, Day 7 and Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- GH Broca-Cochin-Hôtel-Dieu CIC 1417 Cochin-Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided